CLINICAL TRIAL: NCT06659835
Title: Amino Acid Effluent Loss During Continuous Renal Replacement Therapy: an Explorative Non-interventional Pilot Study
Brief Title: Amino Acid Loss During Continuous Renal Replacement Therapy
Acronym: DIAMINO
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Arabella Fischer, MD, Principal investigator, Medical University of Vienna
Other Study IDs: 2149/2023
Record Dates: First submitted 2024-06-30; First posted 2024-10-26 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Renal Insufficiency; Kidney Failure
Keywords: amino acid; continuous renal replacement therapy; effluent loss
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, urine, effluent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CRRT group: intensive care patients with continuous renal replacement therapy
- non-CRRT group: intensive care patients without renal replacement therapy

SUMMARY:
The goal of this observational study is to learn about amino acid loss during continuous renal replacement therapy and plasma amino acid levels in intensive care patients. The main questions it aims to answer are:

What amount of amino acids is lost over the duration of continuous renal replacement therapy? How do amino acid plasma concentrations change over time in patients with and without continuous renal replacement therapy?

Amino acid concentrations will be measured in the effluent and in the plasma of patients receiving continuous renal replacement therapy as part of their regular medical care. In addition, plasma concentrations of amino acids will be studied in patients without renal replacement therapy.

DETAILED DESCRIPTION:
In order to quantify the amount of amino acids lost via the continuous renal replacement (CRRT) machine, it is warranted to measure amino acid concentrations in the blood and effluent over the entire treatment period.

To this end, 20 intensive care patients will be examined throughout the entire duration of CRRT as part of this exploratory non-interventional study. Additionally, 10 intensive care patients without renal replacement therapy will be enrolled. In the CRRT-group amino acid loss through the effluent will be measured at different time points. Amino acid plasma concentrations will be determined in both groups. Amino acid urine concentration, nitrogen balance, as well as blood urea nitrogen, creatinine and albumin in the plasma will be measured as secondary outcome parameters. Additionally, observations regarding nutritional status and mobility (indirect calorimetry, bioimpedance analysis, ultrasound muscle and adipose tissue thickness, strength and mobility scoring) will be analyzed as exploratory secondary outcomes.

Duration of CRRT, length of intensive care and hospital stay as well as mortality will be monitored.

High-performance liquid chromatography fluorescence as well as liquid chromatography-mass spectrometry will be performed to measure amino acid concentrations in plasma, effluent and urine.

To answer the primary research question, change in amino acid plasma concentrations and effluent loss between treatment start and day 4 of continuous renal replacement therapy will be analysed using a two-sided Wilcoxon signed rank test.

ELIGIBILITY:
Inclusion criteria:

* Postoperative ICU patients
* Age ≥ 18 years
* Patients on enteral or/and parenteral nutrition given according to internal standard operating procedure

A) CRRT group:

- CRRT treatment planned; all types of CRRT (continuous veno-venous hemodialysis (CVVHD), continuous veno-venous hemodiafiltration (CVVHDF), continuous veno-venous hemofiltration (CVVH))

B)Non-CRRT group:

* no current or previous (<30 days) continuous or intermittent RRT
* no chronic kidney disease stage G3-G5

Exclusion criteria:

* Preoperative intensive care patients
* Patients with liver cirrhosis stage 1-3 according to the Child-Pugh classification
* Patients with acute liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll 30 intensive care patients: 20 patients receiving continuous renal replacement therapy and 10 patients without renal replacement therapy. The study will be carried out at the Medical University of Vienna at a 16-bed intensive care unit admitting patients after cardiothoracic and major vascular surgery.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Amino acid effluent loss | CRRT start, day 4 of continuous renal replacement therapy
  Change of effluent loss of amino acids from start of continuous renal replacement therapy to day 4
Amino acid plasma concentration CRRT group | day 0, day 4 of continuous renal replacement therapy
  Change of plasma concentration of amino acids from start of continuous renal replacement therapy to day 4
Amino acid plasma concentration non-CRRT group | preoperative day/enrollment to postoperative day 4
  Change of plasma concentration of amino acids from the preoperative day to postoperative day 4 or to the last measurement at the intensive care unit, whichever is earlier

SECONDARY OUTCOMES:
Time course of effluent loss of amino acids over all measured time points | duration of continuous renal replacement therapy, maximum 30 days
  Time course of effluent loss of amino acids over all measured time points
Time course of plasma concentration of amino acids over all measured time points | preoperative if recruited preoperatively, duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Time course of plasma concentration of amino acids over all measured time points
Urine concentration of amino acids over treatment period | preoperative if recruited preoperatively, duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Urine concentration of amino acids over treatment period
Nitrogen balance | duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Nitrogen balance over treatment period
Blood urea nitrogen | preoperative if recruited preoperatively, duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Blood urea nitrogen over treatment period
Creatinine | preoperative if recruited preoperatively, duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Creatinine in blood, effluent, urine over treatment period
Albumin | preoperative if recruited preoperatively, duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Albumin in blood, effluent, urine over treatment period
Total protein | preoperative if recruited preoperatively, duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Total protein in blood, effluent urine over treatment period
Vitamins | duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Vitamins (Vitamin B12, folate) in blood, effluent, urine over treatment period
Trace elements | duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Trace elements (iron, iodide) in blood, effluent, urine over treatment period
Indirect Calorimetry | duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Indirect calorimetry over treatment period
Bioimpedance analysis | preoperative if recruited preoperatively, duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  Bioimpedance analysis over treatment period
Ultrasound Muscle and Adipose Tissue Thickness | preoperative if recruited preoperatively, duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  ultrasound to measure muscle and adipose tissue thickness over treatment period
Muscle Strength | duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  muscle strength assessment (Medical Research Council Scale for Muscle Strength) over treatment period
Mobility | duration of continuous renal replacement therapy (CRRT group) or length of ICU stay (non CRRT-group), maximum 30 days
  mobility assessment (Surgical Intensive Care Unit Optimal Mobilisation Score) over treatment period
Duration of Continuous Renal Replacement Therapy | duration of Continuous Renal Replacement Therapy (CRRT group), through study completion on average 10 days
  duration of Continuous Renal Replacement Therapy
Length of stay | length of ICU and hospital stay, through study completion maximum 1 year
  Length of ICU stay
Mortality | length of ICU and hospital stay, through study completion maximum 1 year
  mortality during ICU and hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Yadavalli, Dr., Principal Investigator — Medical University of Vienna; Arabella Fischer, Dr., Principal Investigator — Medical University of Vienna; Andrea Laßnigg, Prof., Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maxvold NJ, Smoyer WE, Custer JR, Bunchman TE. Amino acid loss and nitrogen balance in critically ill children with acute renal failure: a prospective comparison between classic hemofiltration and hemofiltration with dialysis. Crit Care Med. 2000 Apr;28(4):1161-5. doi: 10.1097/00003246-200004000-00041. PMID 10809299
- [Background] Kihara M, Ikeda Y, Fujita H, Miura M, Masumori S, Tamura K, Yabana M, Takagi N, Umemura S, Ishii M. Amino acid losses and nitrogen balance during slow diurnal hemodialysis in critically ill patients with renal failure. Intensive Care Med. 1997 Jan;23(1):110-3. doi: 10.1007/s001340050299. PMID 9037649
- [Background] Berger MM, Shenkin A, Revelly JP, Roberts E, Cayeux MC, Baines M, Chiolero RL. Copper, selenium, zinc, and thiamine balances during continuous venovenous hemodiafiltration in critically ill patients. Am J Clin Nutr. 2004 Aug;80(2):410-6. doi: 10.1093/ajcn/80.2.410. PMID 15277163
- [Background] Stapel SN, de Boer RJ, Thoral PJ, Vervloet MG, Girbes ARJ, Oudemans-van Straaten HM. Amino Acid Loss during Continuous Venovenous Hemofiltration in Critically Ill Patients. Blood Purif. 2019;48(4):321-329. doi: 10.1159/000500998. Epub 2019 Jul 10. PMID 31291614
- [Background] Story DA, Ronco C, Bellomo R. Trace element and vitamin concentrations and losses in critically ill patients treated with continuous venovenous hemofiltration. Crit Care Med. 1999 Jan;27(1):220-3. doi: 10.1097/00003246-199901000-00057. PMID 9934919
- [Background] Sundstrom Rehal M, Liebau F, Tjader I, Norberg A, Rooyackers O, Wernerman J. A supplemental intravenous amino acid infusion sustains a positive protein balance for 24 hours in critically ill patients. Crit Care. 2017 Dec 6;21(1):298. doi: 10.1186/s13054-017-1892-x. PMID 29212550
- [Background] Bellomo R, Tan HK, Bhonagiri S, Gopal I, Seacombe J, Daskalakis M, Boyce N. High protein intake during continuous hemodiafiltration: impact on amino acids and nitrogen balance. Int J Artif Organs. 2002 Apr;25(4):261-8. doi: 10.1177/039139880202500403. PMID 12027135
- [Background] Chua HR, Bellomo R. Nutritional Management of Patients Treated with Continuous Renal Replacement Therapy. Elsevier Inc.; 2013. https://doi.org/10.1016/B978-0-12-391934-2.00037-0
- [Background] Fischer A, Hertwig A, Hahn R, Anwar M, Siebenrock T, Pesta M, Liebau K, Timmermann I, Brugger J, Posch M, Ringl H, Tamandl D, Hiesmayr M; USVALID Collaboration Group. Validation of bedside ultrasound to predict lumbar muscle area in the computed tomography in 200 non-critically ill patients: The USVALID prospective study. Clin Nutr. 2022 Apr;41(4):829-837. doi: 10.1016/j.clnu.2022.01.034. Epub 2022 Feb 11. PMID 35263692
- [Background] Fischer A, Spiegl M, Altmann K, Winkler A, Salamon A, Themessl-Huber M, Mouhieddine M, Strasser EM, Schiferer A, Paternostro-Sluga T, Hiesmayr M. Muscle mass, strength and functional outcomes in critically ill patients after cardiothoracic surgery: does neuromuscular electrical stimulation help? The Catastim 2 randomized controlled trial. Crit Care. 2016 Jan 29;20:30. doi: 10.1186/s13054-016-1199-3. PMID 26825278
- [Background] Kasotakis G, Schmidt U, Perry D, Grosse-Sundrup M, Benjamin J, Ryan C, Tully S, Hirschberg R, Waak K, Velmahos G, Bittner EA, Zafonte R, Cobb JP, Eikermann M. The surgical intensive care unit optimal mobility score predicts mortality and length of stay. Crit Care Med. 2012 Apr;40(4):1122-8. doi: 10.1097/CCM.0b013e3182376e6d. PMID 22067629
- [Background] Jonckheer J, Vergaelen K, Spapen H, Malbrain MLNG, De Waele E. Modification of Nutrition Therapy During Continuous Renal Replacement Therapy in Critically Ill Pediatric Patients: A Narrative Review and Recommendations. Nutr Clin Pract. 2019 Feb;34(1):37-47. doi: 10.1002/ncp.10231. Epub 2018 Dec 20. PMID 30570180
- [Background] Oddoye EA, Margen S. Nitrogen balance studies in humans: long-term effect of high nitrogen intake on nitrogen accretion. J Nutr. 1979 Mar;109(3):363-77. doi: 10.1093/jn/109.3.363. PMID 430238
- [Background] Bernardi MH, Schmidlin D, Ristl R, Heitzinger C, Schiferer A, Neugebauer T, Wrba T, Hiesmayr M, Druml W, Lassnigg A. Serum Creatinine Back-Estimation in Cardiac Surgery Patients: Misclassification of AKI Using Existing Formulae and a Data-Driven Model. Clin J Am Soc Nephrol. 2016 Mar 7;11(3):395-404. doi: 10.2215/CJN.03560315. Epub 2016 Jan 22. PMID 26801479